CLINICAL TRIAL: NCT02674204
Title: Statin Therapy Operates to Prevent (STOP) Heart Disease in Breast Cancer Survivors Trial
Brief Title: STOP Heart Disease in Breast Cancer Survivors Trial
Acronym: STOP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to low accrual
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: California Breast Cancer Research Program (Other)
Responsible Party: Principal Investigator, Marc Goodman, Professor and Director, Cancer Prevention & Control - Department, Cancer Institute, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT2015-12-Goodman-STOP
Record Dates: First submitted 2016-01-21; First posted 2016-02-04 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer; Heart Disease; Cardiotoxicity; Myocardial Dysfunction
Keywords: Statin therapy; trastuzumab
MeSH Terms: conditions — Breast Neoplasms; Heart Diseases; Cardiotoxicity | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Agent (Experimental): One atorvastatin 20 mg oral capsule per day
  Interventions: Drug: Atorvastatin
- Control (Placebo Comparator): One matching placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin calcium, a synthetic lipid-lowering agent, is an inhibitor of 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase. This enzyme catalyzes the conversion of HMG-CoA to mevalonate, an early and rate-limiting step in cholesterol biosynthesis.
  Other Names: Lipitor; Atorvastatin calcium
  Arms: Study Agent
Drug: Placebo — A substance that has no therapeutic effect, and will be used as a control in testing the study agent.
  Arms: Control

SUMMARY:
The purpose of this study is to to examine the effects of atorvastatin, a type of statin, on changes to the heart among women undergoing breast cancer treatment. Atorvastatin may reduce or eliminate the harmful effects of chemotherapy treatment to the heart tissue of breast cancer patients.

DETAILED DESCRIPTION:
This is a placebo-controlled study. It will compare the effects of atorvastatin against the effects of a placebo (an inactive substance, such as, a sugar pill) on changes to the heart before and during breast cancer treatment. Participants will be in the study for approximately a year and a half, and the study will enroll up to 60 patients. During that time, there will be six visits that may coincide with standard of care visits. Participants will also receive telephone calls from study staff during the study intervention and a follow-up phase to check-in with them.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with newly diagnosed stage 1-3 breast cancer
* Histologically confirmed HER2, ER, and PR status
* Recommended to undergo trastuzumab treatment, with or without anthracycline. Patients will be eligible for up to 3 weeks after starting treatment.
* Age minimum 18 years
* Able and willing to read, understand, and sign an informed consent form (ICF) and medical release form
* Willing and able to comply with trial protocol and follow-up
* ECOG performance status 0-1 (Karnofsky ≥ 70%)

Exclusion Criteria:

* Prior use of statin medication within the past year
* Not using statin medication but is eligible for statin therapy based on the 2013 ACC/AHA guidelines (LDL cholesterol >190, or LDL <190 and ASCVD risk >7.5%; http://tools.acc.org/ASCVD-Risk-Estimator/) and is > 50 years old; or is eligible for statin therapy based on the 2013 ACC/AHA guidelines and is 40-50 years old and wishes to be placed on statin therapy
* History of adverse effects, intolerance, or allergic reactions attributed to statin medication
* Current use of gemfibrozil, cyclosporine, clarithromycin, itraconazole, erythromycin, the hepatitis C protease inhibitor telaprevir, HIV protease inhibitors, colchicine, or red yeast rice
* Current use of any other investigational agent
* Pregnant or intention to get pregnant during the next 18 months. Pregnant women are excluded from this study because atorvastatin is a lipid-lowering agent with the potential for teratogenic or abortifacient effects, and MRI is contraindicated in pregnant women.
* History of diabetes, severe lung disease, renal disease (creatinine > 1.8 mg/dL or CrCl ≤ 50 mL/min), or hepatic disease (AST and ALT > 3 times upper normal limits)
* Abnormal baseline echocardiogram or cardiac MRI (detection of congenital heart disease; ischemic heart disease; moderate or severe valvular heart disease; cardiomyopathy; EF < 55%)
* Previously known or diagnosed heart disease (e.g. congenital; valvular; coronary artery disease; history of myocardial infarction or acute coronary syndrome; cardiomyopathy, including infiltrative, hypertensive, hypertrophic, dilated, constrictive pericarditis, or other cardiomyopathy)
* Left ventricular dysfunction (EF < 55%)
* Prior non-cardiac illness with an estimated life expectancy < 4 years
* Known active infection with HIV
* Allergy or contraindication to MRI testing, including claustrophobia, metallic parts in body the prohibiting MRI, prior gadolinium contrast reaction, or uncontrolled moderate hypertension (sitting blood pressure >160/95 mm Hg with measurements recorded on at least 2 occasions).
* Has metallic breast expanders in place at the time of screening
* Concurrent illness which in the opinion of the investigators would compromise either the patient or the integrity of the data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Goodman, PhD, Principal Investigator — Cedars-Sinal Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Agent | Control
Started | 1 | 1
Completed | 0 | 1
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Agent | Control | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Circumferential Strain (GCS) Measured by Cardiac MRI (CMRI)
Time Frame: baseline to 12 months post initiation of statin intervention
Population: As accrual fell well below target, change in global circumferential strain (GCS) measured by Cardiac MRI (CMRI) was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Global Longitudinal Strain as Measured by CMRI
Time Frame: Baseline to 12 months of follow-up
Population: As accrual fell well below target, change in global longitudinal strain as measured by CMRI was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Peak Left Ventricular Twist as Measured by CMRI
Time Frame: Baseline to 12 months of follow-up
Population: As accrual fell well below target, change in peak left ventricular twist as measured by CMRI was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Peak Left Ventricular Torsion as Measured by CMRI
Time Frame: Baseline to 12 months of follow-up
Population: As accrual fell well below target, change in peak left ventricular torsion as measured by CMRI was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Left Ventricular Untwisting Rate as Measured by CMRI
Time Frame: Baseline to 12 months of follow-up
Population: As accrual fell well below target, change in left ventricular untwisting rate as measured by CMRI was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Left Ventricular Ejection Fraction as Measured by CMRI
Time Frame: Baseline to 12 months of follow-up
Population: As accrual fell well below target, change in left ventricular ejection fraction as measured by CMRI was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Left Ventricular End Diastolic Volume as Measured by CMRI
Time Frame: Baseline to 12 months of follow-up
Population: As accrual fell well below target, change in left ventricular end diastolic volume as measured by CMRI was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Left Ventricular End Systolic Volume as Measured by CMRI
Time Frame: Baseline to 12 months of follow-up
Population: As accrual fell well below target, change in left ventricular end systolic volume as measured by CMRI was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Cardiac Output as Measured by CMRI
Time Frame: Baseline to 12 months of follow-up
Population: As accrual fell well below target, change in cardiac output as measured by CMRI was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Left Ventricular Mass as Measured by CMRI
Time Frame: Baseline to 12 months of follow-up
Population: As accrual fell well below target, change in left ventricular mass as measured by CMRI was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Left Ventricular Concentricity as Measured by CMRI
Time Frame: Baseline to 12 months of follow-up
Population: As accrual fell well below target, change in left ventricular concentricity as measured by CMRI was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Native T1 as Measured by CMRI
Time Frame: Baseline to 12 months of follow-up
Population: As accrual fell well below target, change in native T1 as measured by CMRI was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change in Post Contrast T1 as Measured by CMRI
Time Frame: Baseline to 12 months of follow-up
Population: As accrual fell well below target, change in post contrast T1 as measured by CMRI was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in Extracellular Volume as Measured by CMRI
Time Frame: Baseline to 12 months of follow-up
Population: As accrual fell well below target, change in extracellular volume as measured by CMRI was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change in Native T2 as Measured by CMRI
Time Frame: Baseline to 12 months of follow-up
Population: As accrual fell well below target, change in native T2 as measured by CMRI was not calculated.
Arm/Group | Study Agent | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 12-month intervention period and within 30 days of the last administration of the study drug.
Description: Regular investigator assessment, regular laboratory testing, self-reporting.
Arm/Group | Study Agent | Control
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Agent (N=1) | Control (N=1)
colitis (Gastrointestinal disorders) | 0 | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Agent (N=1) | Control (N=1)
alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
abdominal cramping (Gastrointestinal disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)
pain (General disorders) | 0 (0) | 1 (1)
hot flashes (Reproductive system and breast disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 1 (2)
mood changes (Psychiatric disorders) | 0 (0) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
vitamin D deficiency (General disorders) | 0 (0) | 1 (1)
osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
somnolence (Nervous system disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Accrual fell well below target. Two subjects were randomized to the study and one subject completed the study. Outcome measures were not analyzed due to insufficient accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT02674204/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT02674204/ICF_001.pdf